CLINICAL TRIAL: NCT04102982
Title: Shandong Provincial Hospital Affiliated to Shandong University
Brief Title: Microwave Ablation in Combination With Camrelizumab Versus Camrelizumab in Metastatic Non-small-cell Lung Cancer
Acronym: MWA in NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Xin Ye, Head of Section, Shandong Provincial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Shandong PH
Record Dates: First submitted 2019-09-22; First posted 2019-09-25 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: NSCLC Stage IV
Keywords: NSCLC; Camrelizumab; Microwave ablation; Overall survival; Progression free survival; Objective response rate; Safety
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — camrelizumab

STUDY DESIGN:
Intervention Model Description: Arm 1：Patients in the combination group were treated with MWA in the primary tumor followed by camrelizumab with the dose of 200mg on day 1, repeated every 21 days.
  Arm 2：Patients in the camrelizumab group were treated with camrelizumab with the dose of 200mg on day 1, repeated every 21 days.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Microwave ablation plus camrelizumab group (Active Comparator): Patients in the group are treated with Microwave ablation in the primary tumor, followed by camrelizumab.
  Interventions: Other: Camrelizumab plus microwave ablation
- Camrelizumab group (Placebo Comparator): Patients in the group are treated with camrelizumab alone.
  Interventions: Drug: Camrelizumab

INTERVENTIONS:
Drug: Camrelizumab — Patients will be treated with camrelizumab alone.
  Arms: Camrelizumab group
Other: Camrelizumab plus microwave ablation — In the group, microwave ablation will be administrated to the primary tumors, followed by camrelizumab.
  Other Names: Camrelizumab plus MWA
  Arms: Microwave ablation plus camrelizumab group

SUMMARY:
Patients were randomized to microwave ablation plus camrelizumab group or camrelizumab group.

DETAILED DESCRIPTION:
Patients in the camrelizumab group were treated with camrelizumab with the dose of 200mg on day 1, repeated every 21 days.Patients in the combination group were treated with MWA in the primary tumor followed by camrelizumab with the dose of 200mg on day 1, repeated every 21 days.

The primary end point is overall survival. The second end points include progression free survival, objective response rate and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 75 years old
2. Cytologically or pathologically verified non-small cell lung cancer (NSCLC)
3. Patients with distant metastases or postoperative recurrence
4. EGFR or ALK sensitive mutations are negative (all patients, including non-adenocarcinoma patients)
5. At least one line of platinum-based doublet chemotherapy was administrated
6. Eastern Cancer Cooperative Group（ECOG）Performance Status（PS）of 0 to 1
7. At least two measurable tumors (in other words a measurable tumor lesion exclusive primary tumors)
8. Asymptomatic brain metastases or symptomatic brain metastases under control
9. If treated with irradiation，at least one month interval between radiation and randomization 10）Cardiopulmonary function, laboratory test indicators without ablation or chemotherapy contraindications

11) Informed conssent can be obtained 12) Sufficient tissue specimens for PD-L1 or TMB or blood samples were provided (1 week before treatment, 1 week after ablation, and once every two months for immune evaluation) for subsequent analysis

Exclusion Criteria:

1. Mixed lung cancer contains neuroendocrine tumor, small cell lung cancer or sarcoma
2. Suffering from other malignant tumors within five years
3. EGFR, ALK sensitive mutations are positive or unknown
4. ECOG PS≥2
5. Uncontrolled pleural effusion or pericardial effusion
6. Uncontrolled symptomatic brain metastases
7. Previously anti-PD-1, anti-PD-L1, anti-CTLA-4 or Car-T immunotherapy
8. severe interstitial pneumonia with severe diffuse dysfunction
9. Autoimmune diseases require long-term hormone therapy patients
10. Patients required consistent application of prednisone
11. Uncontrolled pulmonary infection or antibiotics stopped within 1 month
12. Acute cardiovascular and cerebrovascular diseases such as acute cerebral infarction and acute coronary syndrome within 1 month
13. Patients during pregnancy or lactation
14. Life expectance of 3 months or less

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-10-31 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | The proportion of Patients achieved complete response or partial response up to 16 weeks
  ORR

SECONDARY OUTCOMES:
Overall survival | From date of randomization until the date of first documented date of death from any cause，assessed up to 24 months
  OS
Progression free survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  OS
Safety | The proportion and grade of patients had adverse events up to 24 months
  The adverse events of both microwave and camrelizumab

CONTACTS AND LOCATIONS:
Overall Officials: Xin Ye, Principal Investigator — Shandong Provincial Hospital
Locations (13):
- China (13):
  - Binzhou Medical University Hospital, Binzhou, Shandong
  - Dezhou People's Hospital, Dezhou, Shandong
  - The Second People's Hospital of Dezhou, Dezhou, Shandong
  - Jinan Military General Hospital, Jinan, Shandong
  - Affliated Hospital of Shandong Academy of Medical Sciences, Jinan, Shandong
  - Shandong Provincial Hospital affliated to Shandong University, Jinan, Shandong
  - Affliated Hospital of Jining Medical University, Jining, Shandong
  - Liaocheng Cancer Hospital, Liaocheng, Shandong
  - Affliated Hospital of Taishan Medical University, Taian, Shandong
  - The People's Liberation Army 88 Hospital, Taian, Shandong
  - Weifang People's Hospital, Weifang, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Tengzhou center of people's hospital, Zaozhuang, Shandong

IPD SHARING:
Plan to Share IPD: No
Principle of confidentiality